CLINICAL TRIAL: NCT00444847
Title: Effect of Repeated Exposure to Compressed Air on Patients With AIDS (Acquired Immunodeficiency Syndrome)
Brief Title: Effect of Repeated Exposures to Compressed Air on Patients With AIDS
Acronym: DANET1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Designed Altobaric Technology, Incorporated (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DANET HIV/AIDS Trial Q050021; FDA Q050021
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2007-03

CONDITIONS: AIDS
Keywords: AIDS; HIV; Hyperbaric Chamber; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Hyperbaric chamber

SUMMARY:
The exposure of human beings to markedly altered environments (ambient pressure and inhaled gas mixtures) has profound effects on their innate immune capacity to effectively combat viral illnesses. This Phase IIA clinical trial examines the effects of an exposure to a 4 atmospheric environment has on HIV-infected humans whose clinical condition has progressed to formal AIDS status.

ELIGIBILITY:
Inclusion Criteria:

* CD4 count <200
* Viral load > 5000

Exclusion Criteria:

* Opportunistic infection
* Concurrent neoplasm (see protocol)
* Immunomodulators
* HIV vaccination
* Investigational HIV drugs (see protocol)
* Pregnant women
* Major organ transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07

PRIMARY OUTCOMES:
1 - Safety
2 - Viral Load measure (blood and intracellular)
3 - CD4/CD8 levels

SECONDARY OUTCOMES:
ADL measurements

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Guthrie, MD, PhD, Principal Investigator — Designed Altobaric Environment Technology; Stephen G Guthrie, MD, PhD, Principal Investigator — Designed Altobaric Environment Technology
Locations (1):
- Detroit Receiving Hospital, Detroit, Michigan, United States